CLINICAL TRIAL: NCT05322694
Title: Multicenter Prospective Cohort Study to Derive and Validate Clinical Decision Rules in Emergency Department Triage to Improve the Care Pathway for Patients With Acute Respiratory Infection or Acute Infectious Diarrhea.
Brief Title: Clinical Decision Rules in the Emergency Department to Improve the Management of Acute Respiratory Infection and Acute Infectious Diarrhea
Status: Completed | Type: Observational
Sponsor: Simon Berthelot (Other)
Collaborators: Meridian Bioscience, Inc. (Industry); Ministère de l'Économie, de la Science et de l'Innovation (Unknown)
Responsible Party: Sponsor-Investigator, Simon Berthelot, Emergency Physician, CHU de Québec-Université Laval; Associate Professor, Faculté de médecine de l'Université Laval, CHU de Quebec-Universite Laval
Organization: CHU de Quebec-Universite Laval (Other)
Other Study IDs: FACS; CRI-2021-02 (Other: CHU de Québec - Université Laval)
Record Dates: First submitted 2022-03-17; First posted 2022-04-12 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Acute Respiratory Infection; Acute Bacterial Diarrhea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasopharyngeal swab samples and rectal swab samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute respiratory infections: Participants will be recruited according to their symptoms when presenting to the emergency room. They can be included either in the acute respiratory infection group or acute infectious diarrhea group or both.
  Immediately after triage, eligible patients will be approached by research personnel (nurse or other professional authorized to perform the sampling and techniques required for the study) and enrolled after consent has been obtained. Once the study procedures are completed, participants will follow the care pathway that they would normally follow without the research project. The results of the clinical decision rule (molecular test and risk stratification tool) will not be disclosed to the treating team or the patient.
- Acute infectious diarrhea: Participants will be recruited according to their symptoms when presenting to the emergency room. They can be included either in the acute respiratory infection group or acute infectious diarrhea group or both.
  Immediately after triage, eligible patients will be approached by research personnel (nurse or other professional authorized to perform the sampling and techniques required for the study) and enrolled after consent has been obtained. Once the study procedures are completed, participants will follow the care pathway that they would normally follow without the research project. The results of the clinical decision rule (molecular test and risk stratification tool) will not be disclosed to the treating team or the patient.

SUMMARY:
Acute respiratory infections (such as influenza-like illness and upper respiratory tract infection) and acute infectious diarrhea are, for the most part, conditions that do not require medical management or specific treatment. Depending on the level of their transmission in the community, however, these diseases place significant clinical and financial burden on the healthcare system, particularly on emergency departments (ED). The investigators propose a prospective multicenter cohort study with which they aim to validate clinical decision rules combining 1) rapid molecular tests and 2) risk stratification tools to identify patients at low risk for complications related to acute respiratory infection and acute infectious diarrhea. The use of these clinical decision rules by nurses in ED triage could allow low-risk patients to be sent directly home for self-treatment without having to see the emergency physician. By eliminating the need for physician assessment, paraclinical testing and prolonged waiting in the ED, these triage-based clinical decision rules could provide a new, safe care pathway for acute respiratory infections and acute infectious diarrhea, reducing the burden on the patient, the healthcare system, and society.

ELIGIBILITY:
Acute Respiratory Infections :

Inclusion Criteria:

1. 18 years of age or older;
2. Able to consent to the study;
3. Reachable by phone;
4. Consent to be reached directly by phone;
5. At least one of the following respiratory symptoms consistent with an acute respiratory infection for 10 days or less, i. Cough and/or ii. Purulent sputum and/or iii. Pharyngeal pain and/or iv. Nasal congestion and/or v. Rhinorrhea and/or vi. Agueusia and/or vii. Anosmia;
6. A triage score of 3 (30 minutes), 4 (60 minutes) or 5 (120 minutes) on the Canadian Triage and Acuity Scale (CTAS);
7. Triaged by the ED nurse and managed according to standard ED care protocols;
8. Resident of Québec;
9. Holder of a Québec health insurance number.

Exclusion Criteria:

1. Cognitive impairment that prevents the patient from reliably answering the risk stratification tool or research questions;
2. Resident of a long-term care facility;
3. Refusal of nasopharyngeal swab.

Acute infectious diarrhea :

Inclusion Criteria:

1. 18 years of age or older;
2. Able to consent to the study;
3. Reachable by phone;
4. Consent to be reached directly by phone;
5. At least three loose or liquid stools over a 24-hour period and for 10 days or less;
6. A triage score of 3 (30 minutes), 4 (60 minutes) or 5 (120 minutes) on the Canadian Triage and Acuity Scale (CTAS);
7. Triaged by the ED nurse and managed according to standard ED care protocols;
8. Resident of Québec.
9. Holder of a Québec health insurance number.

Exclusion Criteria:

1. Known neutropenia (<500 neutrophils);
2. Active inflammatory bowel disease;
3. Anorectal pathology;
4. Recent colonic surgery (< 6 months);
5. Cognitive impairment preventing the patient from reliably answering the risk stratification tool or research questions;
6. Resident of a long-term care facility;
7. Refusal of the rectal swab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited according to their symptoms when presenting to the ED. They can be included in the acute respiratory infection group, the acute infectious diarrhea group or both.
Sampling Method: Non-Probability Sample
Enrollment: 1474 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
7- and 30-day combined incidence of ED returns, hospitalizations, and deaths. | 30 days
  Combined proportion incidence at 7 and 30 days after the initial visit of ED returns, hospitalizations and deaths related to acute respiratory infection or acute infectious diarrhea (obtained from provincial administrative databases).

SECONDARY OUTCOMES:
Incidence proportion of ED returns | 30 days
  Incidence proportion of ED returns at 7 and 30 days after the initial visit.
Incidence of prescribing antiviral medication | 7 days
  Incidence of prescribing antiviral medication (e.g., oseltamivir) at the initial ED visit and at 7 days (telephone follow-up).
Incidence of antibiotic prescribing | 7 days
  Incidence of antibiotic prescribing at initial visit and at 7 days (telephone follow-up).
Incidence of intensive care unit admission | 30 days
  Incidence of intensive care unit admission at 30 days (obtained from provincial administrative database on hospital admissions).
Mean costs of care of the initial ED visit from a health system perspective | 30 days
  Mean costs of the initial ED visit from a health system perspective estimated using time-driven activity-based costing (data obtained from initial visit data collection, electronic medical records and provincial physician billing database).
Mean costs of the disease from the patient perspective | 7 days
  Mean 7-day costs from the patient perspective (obtained from the Cost for Patient Questionnaire - the CoPaQ- administered at telephone follow-up).
Length of stay in the ED | Measured from ED arrival to ED discharge on the initial visit (maximum 120 hours)
  Length of stay in the ED on the initial visit (electronic medical records).
Incidence proportion of hospitalizations | 30 days
  Incidence proportion of hospitalizations at 7 and 30 days after the initial visit.
Incidence proportion of deaths | 30 days
  Incidence proportion of deaths at 7 and 30 days after the initial visit.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Centre hospitalier universitaire de Montréal, Montreal, Quebec
  - Hôpital Général Juif, Montreal, Quebec
  - CHU de Québec - Université Laval, Québec